CLINICAL TRIAL: NCT05679232
Title: Randomized, Controlled, Monocentric, Feasibility Clinical Investigation to Assess the Safety and Preliminary Clinical Performance of a Hydrogel Coating to Reduce Post-surgical Infection After Joint Arthroplasty
Brief Title: Hydrogel Coating to Reduce Post-surgical Infection After Joint Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P01.025.01
Record Dates: First submitted 2022-12-21; First posted 2023-01-10 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Arthritis; Traumatic Arthritis; Avascular Necrosis
MeSH Terms: conditions — Arthritis; Osteonecrosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study requires a blinded evaluator for the assessment of the primary outcome (i.e. radiological signs of failed osseointegration). The investigators and the participating patients are not blinded to treatment allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrogel coating (Experimental): cementless revision hip arthroplasty with hydrogel coating applied on orthopaedic implants' surfaces
  Interventions: Device: Hydrogel coating
- Control (Sham Comparator): cementless revision hip arthroplasty
  Interventions: Procedure: Control

INTERVENTIONS:
Device: Hydrogel coating — hydrogel coating applied to implant's surfaces during cementless hip revision arthroplasty
  Arms: Hydrogel coating
Procedure: Control — standard cementless hip revision arthroplasty
  Arms: Control

SUMMARY:
The goal of this randomized, controlled, monocentric, single-blind, 2-arm, feasibility clinical investigation is to evaluate the safety of MectaShield hydrogel coating and to capture its preliminary clinical performance in the prevention of early peri-prosthetic joint infection (PJI) in patients undergoing cementless revision hip arthroplasty.

The main questions it aims to answer are:

* demonstrate that the hydrogel coating MectaShield does not interfere with primary stability;
* evaluate clinical and functional outcomes, the rate of PJI and possible adverse events.

Participants will undergo cementless revision hip arthroplasty; during surgery MectaShield hydrogel coating is applied on orthopaedic implants' surfaces (femoral stem and, if revised, acetabular cup) as a protective barrier for the prevention of bacterial adhesion. Surgery and follow-up are completed as per local standard practice. Stability will be assessed radiologically, while functional outcomes and PJI will be monitored by HOOS-PS, ASESPIS scores and according to the consensus document presented by European Society of Radiology (ESRa), the European Association of Nuclear Medicine (EANM), the European Bone and Joint Infection Society (EBJIS), and the European Society of Clinical Microbiology and Infectious Diseases (ESCMID). Researchers will compare the results of the treatment group with those from a control group receiving cementless revision hip arthroplasty without the application of MectaShiled hydrogel coating.

DETAILED DESCRIPTION:
Peri-prosthetic joint infection (PJI) is among the first three reasons for joint replacement failure. PJI is a serious condition that may lead to repeated surgical interventions, prolonged hospitalization, high costs, and significant morbidity, although low mortality. To address this concern, antibacterial coating of implants has been proposed, as the adherence of the microorganisms to the implant, forming a biofilm, plays a strategic role in the pathogenesis of PJI. MectaShield (Medacta International SA) is a novel resorbable hydrogel coating intended to be spread on orthopaedic implants' surfaces as a protective barrier for the prevention of PJI. The study aims to evaluate the safety of MectaShield and to capture its preliminary clinical performance in the prevention of early PJI in patients undergoing cementless revision hip arthroplasty.

Patients suitable to receive MectaShield for cementless revision hip arthroplasty will be invited to take part to the study during the preoperative visit. Follow-up is performed after 3 and 12 months. Data collection includes clinical and functional data for preoperative and postoperative assessments, as well as intraoperative details, adverse events and device deficiencies. Patients will be randomized 1:1 in 2 groups:

* Control (no MectaShield)
* MectaShield hydrogel coating (+ antibiotic)

The primary objective is to demonstrate that MectaShield hydrogel coating does not interfere with early primary stability at 3 months of follow-up

Secondary objectives are:

1. To demonstrate that MectaShield does not interfere with primary stability at 12 months of follow-up
2. To evaluate clinical and functional outcomes at 3 and 12 months of follow-up
3. To evaluate the rate of PJI at 3 and 12 months of follow-up
4. To evaluate the occurrence of adverse events and device deficiencies

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent signed by the subject
* Males and females aged over 18 years at time of surgery
* Subjects who are scheduled to receive a conical collarless cementless revision hip arthroplasty, with or without revision of the acetabular cup
* Subjects willing to comply with the pre- and post-operative evaluation schedule

Exclusion Criteria:

* Subjects with one or more medical conditions identified as a contraindication defined by the labelling on any implants used in this study
* Subjects with immune suppressive treatment for organ transplantation, or known allergy to MectaShield hydrogel constituents (Chitlac, Mannitol, Hydroxypropylmethylcellulose, Sodium phosphate dibasic)
* Subjects presenting with progressive local or systemic infection at the time of surgery
* Subjects whose prospects for a recovery to independent mobility would be compromised by known coexistent, medical problems
* Subjects affected by concomitant spine, hip, ankle or contralateral knee pathologies that can affect walking capacity
* Subjects unable to understand and take action
* Subjects undergoing cementless revision hip arthroplasty in emergency interventions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-12-06 (Actual); Primary Completion 2027-03-06 (Estimated); Study Completion 2027-12-06 (Estimated)

PRIMARY OUTCOMES:
Stem subsidence | 3 months follow up
  Radiological measurements of stem subsidence (mm) will be performed in hydrogel coating and control groups, and mean subsidence will be compared

SECONDARY OUTCOMES:
Stem subsidence | 12 months follow up
  Radiological measurements of stem subsidence (mm) will be performed in hydrogel coating and control groups, and mean subsidence will be compared.
Presence of radiolucent zones in the femur | 3 and 12 months follow up
  Presence of radiolucent lines (≥1 mm) in the 7 Gruen zones will be assessed by radiologic assessment.
Cup migration (if revised) | 3 and 12 months follow up
  Radiological measurements will be performed on the Acetabular cup (if revised) to measure cup migration.
Cup orientation (if revised) | 3 and 12 months follow up
  Radiological measurements will be performed on the Acetabular cup (if revised) to measure cup tilt.
Presence of radiolucent lines in the acetabular cup (if revised) | 3 and 12 months follow up
  Radiological measurements will be performed on the Acetabular cup (if revised) to evaluate the presence of radiolucent lines in the 3 DeLee-Charnley zones (≥1mm).
Clinical and functional outcomes | 3 and 12 months follow up
  Evaluation of daily-life activities, measured with the Hip disability and Osteoarthritis Outcome Score - Physical Function Short Form (HOOS-PS) [0 - 100, worst to best].
Signs of infection | 3 and 12 months follow up
  Evaluation of any sign of infection at the site of surgery, measured with the ASESPIS score (acronym for "Additional treatment, Serous discharge, Erythema, Purulent exudate, Separation of deep tissues, Isolation of bacteria, and Stay as inpatient prolonged over 14 days") [0 - >40, best to worst].
occurrence of PJI | up to 12 months
  The occurrence of PJI is assessed with the diagnostic flowchart proposed by the consensus document issued by the European Society of Radiology (ESRa), the European Association of Nuclear Medicine (EANM), the European Bone and Joint Infection Society (EBJIS), and the European Society of Clinical Microbiology and Infectious Diseases (ESCMID).
Peri-operative and postoperative adverse events and device deficiencies. | up to 12 months
  Monitoring of any peri-operative and postoperative adverse events and device deficiencies.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Dominkus, Prof. Dr., Principal Investigator — Orthopädisches Spital Speising GmbH
Locations (1):
- Orthopädisches Spital Speising GmbH, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No